CLINICAL TRIAL: NCT02983019
Title: Non-interventional Study: Treatment of Influenza in Routine Clinical Practice (FLU-EE)
Brief Title: Treatment of Influenza in Routine Clinical Practice
Acronym: FLU-EE
Status: Completed | Type: Observational
Sponsor: Nearmedic Plus LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: ISIM-LCR
Record Dates: First submitted 2016-11-24; First posted 2016-12-06 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Influenza; Acute Upper Respiratory Infection
Keywords: influenza; flu; acute respiratory viral infection; ARVI; acute upper respiratory infection; AURI
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Therapy with interferons' inducers: Therapy according to routine practice (including Kagocel) Groups will be splitted during the final data analysis
  Interventions: Drug: Kagocel
- Therapy without interferons' inducers: Therapy according to routine practice Groups will be splitted during the final data analysis

INTERVENTIONS:
Drug: Kagocel — Investigators could prescribe other drugs in frame of routine clinical practice
  Groups: Therapy with interferons' inducers

SUMMARY:
This study evaluates the statistics of influenza and acute respiratory viral infections (ARVI) management in outpatient sites in Russia, Armenia, Moldova and Georgia (epidemiology: disease severity and bacterial exacerbations; patients demography; treatment duration and timelines; safety; quality of treatment) in routine clinical practice with focus on drug therapy and usage of interferons' inducers.

DETAILED DESCRIPTION:
This non-interventional study covers more than 15000 patients from outpatient sites in Russia, Armenia, Moldova and Georgia.

Influenza and acute respiratory viral infections (ARVI) diagnosis validate according to "World Health Organization (WHO) Guidelines for Pharmacological Management of Pandemic Influenza A (H1N1) 2009 and other Influenza Viruses". All patients' examinations are carried out according to the local routine clinical practice and local and international standards of care.

The following data will be collected and analyzed after the end of treatment:

* demography
* disease severity
* body temperature
* chills and fever (no/mild/severe)
* weakness (no/mild/severe)
* muscle or joint pain (no/mild/severe)
* rhinitis (yes/no)
* throat irritation (no/mild/severe)
* headache (no/mild/severe)
* cough (no/mild/severe)
* conjunctivitis (no/mild/severe)
* timelines: disease onset, first visit to physician, start of treatment
* therapy (drug name, dose, with focus on interferons' inducers)
* bacterial exacerbations (yes/no)
* therapy of bacterial exacerbations (drug name)
* adverse events
* results of treatment satisfaction questionnaire for medication (TSQM-9), if completed by patient

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years old,
* patients diagnosed with influenza or influenza-like illness caused by a different type of virus,
* patients to whom anti-flu treatment administered,
* patients who have signed informed consent for management of their personal data.

Exclusion Criteria:

* no exclusion criteria except participating in a current clinical trial because of non-interventional sudy design

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with confirmed diagnosis of influenza or influenza-like illness caused by a different type of virus which are on anti-flu therapy
Sampling Method: Non-Probability Sample
Enrollment: 18946 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The socio-demographic data and symptoms of disease in the joint population of patients with influenza and influenza-like illness caused by different types of viruses | up to 14 days
  socio-demographic data, symptoms of disease
The treatment description: names of drugs, dose, time of administration with regards to disease onset ("early" - from 1 to 3 days of symptoms; "late" - 4 or more days of symptoms) | up to 14 days
The efficacy (yes or no) of the treatment schemas with regards to severity of disease (mild, moderate, severe) | up to 14 days
Frequency of influenza complications with antibacterial drugs administration requirement | up to 14 days

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events (AE) with regards to type and severity of AE (mild, moderate, severe; according to physician's opinion) | up to 14 days
Anti-influenza treatment schemas satisfaction rate according to TSQM-9 questionnaire (if completed by patient) | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Sitnikov, Professor, Principal Investigator — Yaroslavl State Medical University
Locations (4):
- Yerevan State Medical University after M. Heratsi, Yerevan, Armenia
- Vl.Bakhutashvili Institute of Medical Biotechnology of Tbilisi State Medical University, Tbilisi, Georgia
- State University of Medicine and Pharmacy Nicolae Testemitanu, Chisinau, Moldova
- Kazan State Medical University, Kazan', Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fazylov VK, Sitnikov IG, Silina EV, Shevchenko SB, Mozhina LN, Zamyatina LL, Yeganyan GA, Groppa LG, Korsantia BM. [Treatment for acute respiratory viral infection and influenza in daily clinical practice: Results of the multicenter international observational FLU-EE study]. Ter Arkh. 2016;88(11):68-75. doi: 10.17116/terarkh2016881168-75. Russian. PMID 28005034